CLINICAL TRIAL: NCT03695133
Title: Effects of Nursing Care Interventions According to Integrative Nursing and Omaha System in Elderly Women Feeling Loneliness: Study Protocol for a Randomized Controlled Trial
Brief Title: Nursing Care Interventions According to Integrative Nursing and Omaha System in Elderly Women Feeling Loneliness
Acronym: INOSEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Aysegul Ilgaz, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Loneliness
Keywords: loneliness; elderly; integrative nursing; omaha system

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): 1. Group-based interventions Group-based interventions include physical activity, sightseeing, picnics, theater, cinema, group educations.
  2. Individual interventions Individual interventions include interventions in the Omaha System Nursing Interventions Scheme that is specific to health problems of elderly women.
  Interventions: Behavioral: Group-based interventions
- control group (No Intervention): The control group will not take any intervention, the post-tests will be collected at the end of 12 weeks.

INTERVENTIONS:
Behavioral: Group-based interventions — 1. Group-based interventions Elderly women will have a walk for physical activity for 12 weeks, three days a week. It is planned that each of the sightseeing, picnic, theater and cinema activities will be done twice. The topics that elderly women need most for group educations will be determined. Group educations will be held once every four weeks approximately three hours.
  2. Individual interventions After the pre-tests are applied to the women in the intervention group, the home environment and the individual's health problems will be assessed, interventions will be implemented and the results will be evaluated during home visits at online. During the home visit to the elderly women and twelve-week intervention period, each woman will meet four times and initiatives will be implemented.
  Other Names: individual interventions
  Arms: intervention group

SUMMARY:
Objectives: The present study investigates the effects of nursing care interventions on the physical, psychological, social and spiritual health of the elderly women with high level of loneliness according to the principles of integrative nursing and Omaha System.

Methods: This study protocol describes a randomised controlled trial with to parallel group design. After the level of loneliness of elderly women will be determined by the Loneliness Scale for the Elderly in the Family Health Center, women with high levels of loneliness will be randomly assigned to the intervention and control group. Nursing care interventions consisting of group-based (sightseeing, picnics, theater, cinema) and individual according to Integrative Nursing and Omaha System. Elderly women who feel loneliness will continue for 12 weeks. Pre-tests and post-tests will be completed during home visits made by the researchers.

Discussion: This study will provide evidence regarding the effectiveness of nursing care interventions that include the comprehensive (physical, psychological, social and spiritual) evaluation of their health, and contribute to provide care in terms of Integrative Nursing and Omaha System.

ELIGIBILITY:
Inclusion Criteria:

* to be independent according to the Katz Daily Activities Activity Scale;
* no problem in physical activity with the suggestion of the doctor in Family Health Center;
* living alone or with family;
* good cognitive state (place, time and person orientation) with the suggestion of the doctor; - the willingness to participate in the study

Exclusion Criteria:

* to live in any elderly care center or nursing home;
* to be semi-dependent and dependent according to the Katz Daily Activities Activity Scale
* to have a psychiatric disorder.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — to feel very lonely and very lonely according to the Loneliness Scale for the Elderly
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Loneliness Scale for the Elderly | 12 weeks
  The loneliness scale for the elderly was developed to determine the sense of loneliness. The two subscales in the scale are: emotional and social loneliness subscales. There are 11 items in the binary Likert type scale. Minumum and maximum scores are 0 and 22 points, respectively. The total score is obtained by collecting the scores from the subscales. Loneliness can be divided into four levels according to the score. "0-4 scores" do not feel loneliness, "5-14 scores" acceptable loneliness, "15-18 scores" feeling very loneliness and "19-22 scores" feeling very lonely. Levels increase the level of loneliness.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | 12 weeks
  There are 7 questions in the short form of the questionnaire. This measure assesses the types of intensity of physical activity. The items in the short form were structured to provide separate scores on walking, moderate-intensity and vigorous-intensity activity. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities. Standard MET values for activities were established. Total Work MET-minutes/week =sum of Walking+Moderate+Vigorous MET-minutes/week scores at work. The score obtained is classified as non-physical activity (MET-600 energy level), insufficient physical activity level (MET = energy level between 600-3000) and adequate physical activity level (MET ≥ 3000 energy level).
Health Status Perception Scale | 12 weeks
  In order to determine the perception of health status, it is questioned how the individual evaluates his / her health now. Very good (1), good (2), bad (3) and very bad (4) options on the scale, the lowest score is 4, the highest score is 1.
Social Inclusion Scale | 12 weeks
  Social inclusion scale evaluates that whether having the opportunities and resources to participate fully in economic, social and cultural life and to enjoy a standard of wellbeing that is considered normal in the society in which we live or not. There are three subscales in the Lİkert type scale, consisting of 18 items: Social Isolation, Social Relations and Social Acceptance. The lowest score is 1 and the highest score is 72. As the score obtained from the scale increases, social inclusion is increasing.
Multidimensional Scale of Perceived Social Support | 12 weeks
  There are 12 items on the scale evaluating the adequacy of social support. In this scale, there are three sub-dimensions: family, friend and special human support. The sum of the obtained scores is collected separately for each subgroup and the sum of these groups gives the total score of the scale. The lowest score is 4 and the highest score is 28 from subscales. The lowest score is 12 and the highest score is 84 from total scale. The higher the score, the higher the perceived social support.
Well-being Index | 12 weeks
  This index evaluates the general emotional state. There are five items in the six-point likert type index. Questions that ask individuals how they often feel in the last two weeks are scored from 0 to 5. In this index, the points taken from the questions are collected and multiplied by four to 0-100 points. As the score from the index increases, it means that the emotional situation is good.
Healthy Life Style Behavior Scale II (spiritual development sub-scale) | 12 weeks
  It was developed to measure health promotion behaviors of individuals. The scale consists of 52 items and six factors (health responsibility, physical activity, nutrition, spiritual development, interpersonal relations and stress management). In this study, spiritual development subscale was used. Likert type scale is scored from 1 to 4. The lowest nine scores from the spiritual development subscale and the highest 36 points are taken. Increasing the score from the scale indicates that the spiritual development is good.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül ILGAZ, Principal Investigator — Research Assistant
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I want to share a study protocol with other researchers.
Supporting Information: Study Protocol
Time Frame: one year
URL: https://pubmed.ncbi.nlm.nih.gov/33317377/

REFERENCES:
- [Derived] Ilgaz A, Gozum S. Effectiveness of INOSEL program consisting of Integrative Nursing and Omaha System for older women feeling loneliness: a randomised controlled trial. Aging Clin Exp Res. 2023 Nov;35(11):2769-2781. doi: 10.1007/s40520-023-02559-9. Epub 2023 Sep 28. PMID 37759148